CLINICAL TRIAL: NCT02156050
Title: Utilisation du Dispositif BBloo® Pour le Traitement de l'ictère néonatal : Satisfaction Des Parents et Des Personnels Soignants
Brief Title: Use of a New Phototherapy Device (BBloo®) for the Treatment of Hyperbilirubinemia in the Newborn Infant
Acronym: ICT-O2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Pédiatrique des Groupes d'Acuueil et de Recherche (Other)
Collaborators: Hopital Antoine Beclere (Other); Bicetre Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICT-O2
Record Dates: First submitted 2014-05-16; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OBLOO device (MEDIPREMA) (Active Comparator): two sessions of 4 hours Phototherapy treatment
  Interventions: Device: two sessions of 4 hours Phototherapy treatment
- BBLOO Device (MEDIPREMA) (Experimental): two sessions of 4 hours Phototherapy treatment
  Interventions: Device: two sessions of 4 hours Phototherapy treatment

INTERVENTIONS:
Device: two sessions of 4 hours Phototherapy treatment — two sessions of 4 hours Phototherapy treatment

SUMMARY:
Jaundice occurs in most newborn infants. Most jaundice is benign, but because of the potential toxicity of bilirubin, newborn infants must be monitored to identify those who might develop severe hyperbilirubinemia an, in rare cases, acute bilirubin encephalopathy or kernicterus. Jaundice is a commonly observed, usually harmless condition in newborn infants during the first week after birth. However, in some babies the amount of bilirubin pigment can increase to dangerous levels and require treatment. Treatment of jaundice in newborn infants is done by placing them under phototherapy, a process of exposing their skin to light of a specific wavelength band. Fluorescent tubes or halogen lamps have been used as light sources for phototherapy for many years. A light-emitting diode (LED) is a newer type of light source which is power efficient, has a longer life and is portable with low heat production. Several technologies and devices are developed around this LED and specially a compact system.

The purpose of this study is to evaluate efficacity of LED phototherapy by comparing with conventional phototherapy (non-LED) and satisfaction of the parents and the professional staff about comfort of this new technology. The newborn infant is placed in a sleeper with the device B' bloo ® which maintains him in position (lap or dorsal) allowing to pass the blue light. This one is generated by the module LED and transmitted in the braid of optical fibers which takes place directly on the mattress of the cradle in which is placed the patient usually.

The device is endowed with an hour counter to schedule the time of treatment. The energy illumination varies between 3 and 4 mW / cm ² for an average 3,6 mW / cm ².

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants ≥ 38 gestation weeks without or with risk factors of severe icterus (G6PD or pyruvate-kinase deficiency, red blood cells membrane defects, hemoglobinopathies, cephalohematoma or significant bruising, decreased breastfeeding)
* newborn at 35 and 38 gestation weeks without risk factor of severe icterus (qs)
* hyperbilirubinemia to deal according to the curves of indication of phototherapy of the APP on 2004
* no opposition of parents

Exclusion Criteria:

* opposition of parents
* newborn infants less than 33 weeks
* newborn infants at 35 or more weeks of gestation with risk factors of severe icterus
* Jaundice in first 12 hours
* Hyperbilirubinemia > 340 µmol/L whatever is the age

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
EDIN Scale | base line, 60minutes, 240minutes
  EDIN scale will be measured 3 times during phototherapy treatment (base line, at 1 hour and at 4 Hour)

SECONDARY OUTCOMES:
Evaluation of Blood Bilirubin level | base line, at 12 hour and at 24 hour
  blood bilirubin concentration will be measured 3 times during phototherapy treatment (base line, at 12 hour and at 24 Hour)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - hopital Antoine Béclère, Clamart
  - Bicetre Hospital, Le Kremlin-Bicêtre